CLINICAL TRIAL: NCT01593657
Title: Mindful Movement and Breathing to Improve Outcomes of Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00019838; CCCWFU 01112 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-05-02; First posted 2012-05-08 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Gynecologic Malignancy; Abdominal Surgery by Laparotomy; Pain; Psychological Distress; Lung Function; Surgical Complications
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Movement and Breathing program (Experimental): Mindful Movement and Breathing program implemented in a hospital room or clinic room three times by a yoga instructor: prior to surgery, one day and two days after surgery.
  Interventions: Other: Mindful Movement and Breathing program; Other: Questionnaire administration; Procedure: The Observer Mobility Scale; Procedure: Volumetric Incentive Spirometry

INTERVENTIONS:
Other: Mindful Movement and Breathing program — Participate Mindful Movement and Breathing program with an experienced yoga instructor. All movements can be done while in a bed (e.g. turning head, shrugging shoulders, bending knees, etc). Each session lasts approximately 15 minutes.
Other: Questionnaire administration — Collected at baseline (before surgery), before and after each YST session, and at follow-up (two days after surgery).
Procedure: The Observer Mobility Scale — Conducted by nurse and study coordinator prior to surgery and two days after surgery to assess mobility. Will ask patient to turn, sit, stand and walk as they are able.
Procedure: Volumetric Incentive Spirometry — Conducted twice before and after each Mindful Movement and Breathing program to measure lung function. Mean of the two readings used.

SUMMARY:
The purpose of this clinical trial is to understand if women undergoing surgery for a suspected gynecologic malignancy are interested in participating in a Mindful Movement and Breathing program and what the effects of this program are on women and the surgery-related symptoms they experience. Mindful Movement and Breathing programs may be effective for easing distress, post-surgical pain, and other symptoms of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed protocol specific informed consent
* 18 years of age or older
* Scheduled for a major abdominal gynecological surgery to remove a mass that is suspected to be malignant

Exclusion Criteria:

* Unable to read or understand English
* Cognitively impaired and/or cannot complete interviews as judged by the referring physician, nurse, or study staff

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing and evaluating a Mindful Movement and Breathing Program among women undergoing gynecologic surgery for a suspected malignancy (recruitment, retention, adherence, and program evaluation and acceptability rates) | 4-5 days
  The proportion of participants who participated in all YST sessions and those who completed all assessments will be computed and compared to those with incomplete data by demographic characteristics. We will model the relationship between adherence and baseline scores of the measures, as well as change in scores. We will also calculate the proportions and 95% confidence intervals of the items that measure program evaluation and intervention to the Clinical Studies Coordinator, nurses and yoga instructor.

SECONDARY OUTCOMES:
Immediate effects of the Mindful Movement and Breathing program on reducing postsurgical pain, psychological distress and lung function | 4-5 days
  Measured using Immediate Effect Visual Analog Scales (VAS) of pain and distress and percent change in inspiratory capacity as assessed with a Volumetric Incentive Spirometer. Assessed for each measure by day using a paired t-test and overall using a mixed effects model on the pre-post change in the measure over time.
Collect data on measures that will be used to evaluate the efficacy of the Mindful Movement and Breathing program in a future larger randomized controlled trial | 4-5 days
  means and standard deviations of the measures will be calculated to inform sample size calculations for a future study, and to provide descriptive statistics of the sample population.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States